CLINICAL TRIAL: NCT00054522
Title: Calcitriol + Dexamethasone in Early, Recurrent Prostate Cancer Following Local Therapy, A Phase I/II Trial
Brief Title: Calcitriol and Dexamethasone in Treating Patients With Prostate Cancer Who Have Undergone Surgery or Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Donald Trump, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270758; RPCI-RP-0203
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: dexamethasone

SUMMARY:
RATIONALE: Calcitriol may help tumor cells develop into normal cells. Dexamethasone may increase the effectiveness of calcitriol by making tumor cells more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of combining calcitriol with dexamethasone in treating patients with prostate cancer who have undergone surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether calcitriol and dexamethasone can slow the rise in prostate-specific antigen (PSA) levels in patients with early, recurrent prostate cancer after prior radical prostatectomy or radiotherapy.
* Determine the safety of this regimen in these patients.
* Determine the utility of serum PSA in monitoring the therapeutic effect of calcitriol in these patients.

OUTLINE: Patients are stratified according to prior therapy (radical prostatectomy vs radiotherapy).

Patients receive oral calcitriol once daily on days 1-3 alone on week 1. Beginning on week 3, patients receive calcitriol as in week 1 and oral dexamethasone on days 0-4. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 56 patients (28 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate meeting all of the following criteria:

  * Curatively treated with radical prostatectomy OR definitive radiotherapy
  * No signs of clinical recurrence or dissemination of prostate cancer by digital rectal examination without tumor
  * No local recurrence by CT scan or MRI of the pelvis
  * No metastases by bone scan and chest x-ray NOTE: Prior Prostascint scans allowed regardless of results
* At least 3 prostate-specific antigen (PSA) measurements obtained over at least 90 days after radical prostatectomy on post-radiotherapy PSA nadir must be available

  * PSA at least 2 ng/mL after prostatectomy OR at least 4 ng/mL after prior radiotherapy
  * Patients previously treated with radiotherapy must have a PSA clearly rising from lowest value within 6 months after completion of therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 12 months

Hematopoietic

* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN

Renal

* Creatinine less than 1.8 mg/dL
* Phosphorus normal
* No hypercalcemia (albumin-corrected calcium greater than ULN)
* No nephrolithiasis

  * Single episode of renal lithiasis allowed provided episode occurred more than 5 years prior to study

Other

* Fertile patients must use effective double-barrier contraception for at least 1 week before, during, and for at least 2 weeks after study
* No symptomatic pancreatitis
* No uncontrolled diabetes
* No known or suspected inability to comply with study requirements (e.g., abuse of alcohol/drugs or psychotic states)
* Curatively treated condition associated with renal stones (e.g., hyperparathyroidism, bladder dysfunction, or obstructive uropathy) allowed provided patient has been free of stone formation for more than 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for prostate cancer
* At least 24 months since prior chemotherapy for other diseases

Endocrine therapy

* More than 6 months since prior hormonal therapy, including neoadjuvant or adjuvant androgen deprivation therapy (e.g., luteinizing hormone-releasing hormone analogue or antiandrogen)
* No prior androgen deprivation therapy of more than 8 months duration
* No prior hormonal therapy for prostate cancer more than 3 months after definitive local therapy
* No concurrent androgen therapy

Radiotherapy

* See Disease Characteristics
* More than 3 months since prior radiotherapy for locally recurrent prostate cancer
* No concurrent radiotherapy, including for pain control

Surgery

* See Disease Characteristics

Other

* More than 4 weeks since prior investigational drugs
* No concurrent medication known to affect systemic calcium metabolism, including any of the following:

  * More than 400 IU of cholecalciferol supplements
  * More than 500 IU of vitamin A supplements
  * Calcium supplements
  * Fluoride
  * Antiepileptics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-04; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Study Chair — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania